CLINICAL TRIAL: NCT07096206
Title: Natural History and Disease Burden of X-linked Hypohidrotic Ectodermal Dysplasia (XLHED): An Observational, Multicentre, International Study (EdeReaLife)
Brief Title: Characteristics and Impacts of X-linked Hypohidrotic Ectodermal Dysplasia (XLHED) in Boys: An Observational International Study
Acronym: EdeReaLife
Status: Active, not recruiting | Type: Observational
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS16479
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: X-Linked Hypohidrotic Ectodermal Dysplasia (XLHED)
Keywords: Observational study; X-Linked Hypohidrotic Ectodermal Dysplasia; XLHED; EDA null mutation
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, multicentre, international study over a 2-year follow-up period.

The aim of this study is to understand how XLHED affects the lives of young male patients and their families over time. By studying the natural course of the disease and its impact, the study could improve the understanding of the challenges faced by these patients and their families.

DETAILED DESCRIPTION:
XLHED is a rare genetic condition that affects more severely males. The main symptoms are missing or reduced ability to sweat, leading to a risk of dangerous overheating, as well as few or no teeth and sparse hair. This condition can significantly impact the daily lives of patients and their families.

Given the rarity of the disease and the purely descriptive purposes of the study, all eligible patients may be included over a period of approximately 12 months. It is expected to include between 20 and 30 male patients over one year of enrolment in France and Germany.

Statistical analysis: will be descriptive with no hypothesis tested. Questionnaires will be completed by the child's parent at inclusion and at 1 and 2 years after the inclusion data

ELIGIBILITY:
Inclusion Criteria:

* Boy
* Age at inclusion: from birth to the day before the 11th birthday
* XLHED disease that has been diagnosed by:
* genetic testing or
* symptoms (sweating ability, teeth and hair impairment) and genetic diagnosis of the mother

Exclusion Criteria:

* Any previous treatment with ER004 or participation in a clinical trial testing ER004
* Testing for XLHED disease with a negative result

Ages: 0 Years to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Study Population: National expert centres specialized in XLHED in France and Germany
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2026-11-19 (Estimated); Study Completion 2026-11-19 (Estimated)

PRIMARY OUTCOMES:
Age | At inclusion
  mean age
Ectodysplasin A (EDA) characterization of the mutation (null or hypomorphic) | at inclusion
  % of patients
Mean sweat volume (µL) | at inclusion
  mean (µL)
Mean sweat volume (µL) | at one year
  mean (µL)
Mean sweat volume (µL) | at two years
  mean (µL)
Sweat pore density | at inclusion
  % of patients with normal/abnormal sweat pore density
Sweat pore density | at one year
  % of patients with normal/abnormal sweat pore density
Sweat pore density | at two years
  % of patients with normal/abnormal sweat pore density
Dentition problem (anodontia, hypodontia, oligodentia) | at inclusion
  % of patients
Dentition problem (anodontia, hypodontia, oligodentia) | at one year
  % of patients
Dentition problem (anodontia, hypodontia, oligodentia) | at two years
  % of patients
Dry eyes | at inclusion
  % of patients
Dry skin | at inclusion
  % of patients

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) at inclusion | at inclusion
  mean +/- SD of the Global score
PedsQL (parent report) | at inclusion
  mean +/- SD of the Global score

CONTACTS AND LOCATIONS:
Overall Officials: Marlène Guiraud, Study Director — Pierre Fabre Médicament
Locations (2):
- Necker hospital, Paris, France
- Uniklinikum Erlangen, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No